CLINICAL TRIAL: NCT01776892
Title: Collagenase and Needle Aponeurotomy: Single Modality Versus Combination Treatment for Dupuytren's Disease
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dupuytren's 001
Record Dates: First submitted 2013-01-17; First posted 2013-01-28 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Dupuytren Contracture
Keywords: Collagenase; Needle aponeurotomy
MeSH Terms: conditions — Dupuytren Contracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Collagenase and needle aponeurotomy (Experimental): Participants in this arm of the study will be treated once with needle aponeurotomy and up to 3 times at 4 week intervals with collagenase injection.
  Affected Dupuytren's cords will be treated with 1-3 collagenase clostridium histolyticum injections at 4 week intervals, based on clinical response of the contracture. Cords will be treated until motion of the joint is within 0-5 degrees of normal, for up to 3 total injections.
  Percutaneous needle aponeurotomy will be performed using an 18 gauge needle. The needle is inserted through the skin into the Dupuytren's cord. The needle is moved very slowly through the cord until complete rupture of the cord is obtained.
  Interventions: Drug: Collegenase injection; Procedure: Needle aponeurotomy
- Needle aponeurotomy (Active Comparator): Percutaneous needle aponeurotomy will be performed using an 18 gauge needle. The needle is inserted through the skin into the Dupuytren's cord. The needle is moved very slowly through the cord until complete rupture of the cord is obtained. Participant feedback is obtained throughout the procedure to prevent digital nerve or flexor tendon injury. Participants are asked to report Tinel's sign which indicates that the needle is in close proximity to the digital nerve and to report pain with needle advancement which indicates proximity to the flexor tendon.
  Interventions: Procedure: Needle aponeurotomy
- Collagenase injection (Active Comparator): Collagenase clostridium histolyticum will be used to treat participants in this arm of the study. Affected cords will be treated with 1-3 collagenase injections at 4 week intervals, based on clinical response of the contracture. Cords will be treated until motion of the joint is within 0-5 degrees of normal, for up to 3 total injections. Metacarpophalangeal cords will be injected with 0.58mg (10 000 units) of collagenase in 0.25ml of sterile diluent. Proximal interphalangeal cords will be injected with 0.58mg (10 000 units) of collagenase in 0.20ml of sterile diluent.
  Interventions: Drug: Collegenase injection

INTERVENTIONS:
Drug: Collegenase injection — Collagenase clostridium histolyticum will be used to treat participants in this arm of the study. Affected cords will be treated with 1-3 collagenase injections at 4 week intervals, based on clinical response of the contracture. Cords will be treated until motion of the joint is within 0-5 degrees of normal, for up to 3 total injections.
  Metacarpophalangeal cords will be injected with 0.58mg (10 000 units) of collagenase in 0.25ml of sterile diluent. Proximal interphalangeal cords will be injected with 0.58mg (10 000 units) of collagenase in 0.20ml of sterile diluent.
  Other Names: Trade name: Xiaflex.
  Arms: Collagenase and needle aponeurotomy; Collagenase injection
Procedure: Needle aponeurotomy — Percutaneous needle aponeurotomy will be performed using an 18 gauge needle. The needle is inserted through the skin into the Dupuytren's cord. The needle is moved very slowly through the cord until complete rupture of the cord is obtained.
  Arms: Collagenase and needle aponeurotomy; Needle aponeurotomy

SUMMARY:
Dupuytren's disease results in deformity of the hand and this can lead to trouble with daily activities. Treatment traditionally involves cutting out diseased tissue, however this can cause damage to important structures in the hand and results in large scars.

Needle aponeurotomy and collagenase injections are newer treatments that are thought to be safer. These treatments allow quicker return to function. One drawback is that Dupuytren's deformity may return more quickly than when all diseased tissue is surgically cut out.

This research study is designed to compare the effectiveness of needle aponeurotomy and collagenase injection for Dupuytren's disease. This study will determine which procedure gives the best results- either needle aponeurotomy, collagenase injection, or both procedures in combination. Participants will be evaluated to see how they do in the long term.

DETAILED DESCRIPTION:
Dupuytren's disease is a benign proliferative disorder of the palmar fascia. It results in progressive thickening and contracture of fibrous bands on the volar surface of the palm and fingers as a result of excessive myofibroblast activity. Patients develop longitudinal cords which may lead to progressive joint contractures. Dupuytren's disease limits hand function and can diminish quality of life.

The most commonly used technique for treatment is open limited fasciectomy. The cumulative complication rate ranges from 14-67% and includes nerve division (2-5%), infection (4-12%), neurapraxia (0.4-52%), and regional pain syndrome (2-13%). The recurrence rate of Dupuytren's disease after fasciectomy is approximately 50% at 5 years.

Recently, interest in needle aponeurotomy and collagenase clostridium histolyticum injection have increased as alternative treatment modalities for Dupuytren's disease. Both procedures can be performed in an outpatient clinic, have limited downtime, allow earlier return to work, and are associated with significantly fewer serious complications than open fasciectomy. Needle aponeurotomy and collagenase injection are less invasive than fasciectomy, however they are associated with higher rates of disease recurrence.

Numerous studies investigating the effectiveness and safety of needle aponeurotomy and collagenase injection studies have been published. To date, there is no published literature about the use of these techniques in combination for the treatment of Dupuytren's disease. The investigators propose to follow the patient population of a single surgeon performing needle aponeurotomy in combination with collagenase injection to determine the effectiveness of this combination treatment. Patients treated with combination treatment will be compared to patients treated with a single modality- either needle aponeurotomy or collagenase injection.

Patients will be assessed pre and post operatively to evaluate functional status and the degree of joint contracture. Patient satisfaction, adverse events, recurrence, and repeat treatment rates will also be determined.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Metacarpophalangeal joint contracture between 20-100 degrees OR proximal interphalangeal joint contracture between 20-80 degrees
* Positive table top test, defined as the inability to simultaneously place the affected finger and palm flat on a table

Exclusion Criteria:

* Use of an anticoagulant within 7 days before the beginning of the study, excluding aspirin
* Bleeding disorder
* Recent stroke
* Allergy to collagenase
* A chronic muscular, neurologic, or neuromuscular disorder affecting the hands
* Previous treatment of the affected joint within 90 days before the beginning of the study
* Use of a tetracycline derivative within 14 days before the beginning of the study
* Pregnancy
* Breast feeding
* Premenopausal woman, not using contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Degree of joint contracture post treatment | 5 years post treatment
  The degree of the participant's Dupuytren's disease joint contracture after treatment will be measured by a physical therapist at each of the participant's follow up appointments.

SECONDARY OUTCOMES:
Change in joint range of motion | Baseline and 5 years post treatment
  The participant's range of motion in their joint affected by Dupuytren's disease will be measured by a physical therapist prior to treatment and following treatment at each of the participant's follow up appointments.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Morhart, MD MSc, Principal Investigator — Division of Plastic Surgery, Department of Surgery, University of Alberta
Locations (1):
- Royal Alexandra Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Badalamente MA, Hurst LC. Enzyme injection as nonsurgical treatment of Dupuytren's disease. J Hand Surg Am. 2000 Jul;25(4):629-36. doi: 10.1053/jhsu.2000.6918. PMID 10913202
- [Background] Badalamente MA, Hurst LC, Hentz VR. Collagen as a clinical target: nonoperative treatment of Dupuytren's disease. J Hand Surg Am. 2002 Sep;27(5):788-98. doi: 10.1053/jhsu.2002.35299. PMID 12239666
- [Background] Hurst LC, Badalamente MA, Hentz VR, Hotchkiss RN, Kaplan FT, Meals RA, Smith TM, Rodzvilla J; CORD I Study Group. Injectable collagenase clostridium histolyticum for Dupuytren's contracture. N Engl J Med. 2009 Sep 3;361(10):968-79. doi: 10.1056/NEJMoa0810866. PMID 19726771
- [Background] Gilpin D, Coleman S, Hall S, Houston A, Karrasch J, Jones N. Injectable collagenase Clostridium histolyticum: a new nonsurgical treatment for Dupuytren's disease. J Hand Surg Am. 2010 Dec;35(12):2027-38.e1. doi: 10.1016/j.jhsa.2010.08.007. PMID 21134613
- [Background] van Rijssen AL, Ter Linden H, Werker PMN. Five-year results of a randomized clinical trial on treatment in Dupuytren's disease: percutaneous needle fasciotomy versus limited fasciectomy. Plast Reconstr Surg. 2012 Feb;129(2):469-477. doi: 10.1097/PRS.0b013e31823aea95. PMID 21987045